CLINICAL TRIAL: NCT03426436
Title: Evaluation of Synthesized 18-Lead ECG in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nihon Kohden (Industry)
Collaborators: Feinstein Institute for Medical Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-0936
Record Dates: First submitted 2018-02-01; First posted 2018-02-08 (Actual); Results first posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-10

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Masking Description: The cardiologist will be blinded to the type of waveform they are analyzing (synthesized versus actual).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Test (Other): Obtain two consecutive 15-lead ECGs; The first 15-lead ECG will have an additional three electrodes/stickers on the right side of the chest and the second 15-lead ECG will have an additional three electrodes/stickers on the posterior side.
  Interventions: Diagnostic Test: Two consecutive 15-lead ECGs

INTERVENTIONS:
Diagnostic Test: Two consecutive 15-lead ECGs — The 15-lead ECG consists of a traditional 12-lead ECG and an additional three leads on the right side of the body. The first 15-lead ECG will have an additional three electrodes/stickers on the right side of the chest and the second 15-lead ECG will have an additional three electrodes/stickers on the posterior side.

SUMMARY:
This study, sponsored by Nihon Kohden, aims to determine the sensitivity and specificity of synthesized 18-lead electrocardiogram (ECG) in the diagnosis of posterior-lateral and/or right-ventricular ischemia, using actual 18-lead ECG as the gold standard. The synthesized 18-lead ECG calculates six extra leads of information from the standard 12-lead ECG done in the Emergency Department (ED). Nihon Kohden has created synECi18 Technology, which can mathematically synthesize and display the extra leads.

The patient population (n=300) will consist of patients who present to the North Shore University Hospital or Long Island Jewish Medical Center ED with a chief complaint of chest pain, chest pressure, or chest discomfort. These patients will be receiving a standard 12-lead ECG as part of their routine clinical care. Patients with ST-Elevation Myocardial Infarction (STEMI) and a known positive troponin value will be excluded from the study.

Trained ED study technicians will use ECG machines provided by Nihon Kohden to obtain two consecutive 15-lead ECGs. The two 15-lead ECGs are then saved onto the ECG machine.The saved information will later be input into an algorithm to calculate the synthesized 18-leads. The actual 18-leads (composed of the two 15-leads conducted in the ED) will be compared with the synthesized 18-leads produced by the synECi18 technology. A study cardiologists will evaluate the actual 18-lead ECGs and synthesized 18-lead ECGs and determine whether there is posterior-lateral and/or right-sided ventricular ischemia. The cardiologists will be blinded to the type of waveform they are analyzing (synthesized versus actual).

The study will not interfere with patient care or treatment, however, the two 15-lead ECGs done in the ED will be shown to the physician who can determine whether or not to order an official 18-lead ECG in the hospital's electronic medical record system.

It is hypothesized that the synECi18 synthesized 18-lead ECGs will provide high sensitivity and specificity for diagnosing posterior-lateral and/or right-ventricular ischemia, with the actual 18-lead ECGs being used as the reference for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a chief complaint of chest pain or chest discomfort or chest pressure
* Troponin test has been ordered (unknown positive at time of recruitment)
* Subjects are capable of providing informed consent
* English speaking

Exclusion Criteria:

* STEMI patients
* Patients who have not had a troponin test ordered
* Pregnant women
* Patients under 18 years of age
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2019-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timmy Li, PhD, Principal Investigator — Northwell Health
Locations (2):
- United States (2):
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test
Started | 314
Completed (16 subjects excluded from analysis) | 295
Not Completed | 19
Not completed — Incorrect lead placement | 12
Not completed — Withdrawal by Subject | 2
Not completed — Consent issue | 1
Not completed — ECGs not saved | 4

BASELINE CHARACTERISTICS:
Arm/Group | Test
Number analyzed (Participants) | 295
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150
  Male | 145
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 295

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity Agreement Between Synthesized and Actual 18-lead ECGs in the Identification of ST Elevation, ST Depression, and T Wave Inversion
Description: Sensitivity, Specificity, Positive Predictive Value and Negative Predictive Value for comparison of actual 18-lead ECG vs synthesized ECG leads. All measures at 95% confidence Index.
Time Frame: 30 minutes
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Participants: Obtain two consecutive 15-lead ECGs; The first 15-lead ECG will have an additional three electrodes/stickers on the right side of the chest and the second 15-lead ECG will have an additional three electrodes/stickers on the posterior side.
  Two consecutive 15-lead ECGs: The 15-lead ECG consists of a traditional 12-lead ECG and an additional three leads on the right side of the body. The first 15-lead ECG will have an additional three electrodes/stickers on the right side of the chest and the second 15-lead ECG will have an additional three electrodes/stickers on the posterior side.
Arm/Group | All Participants
Number analyzed (Participants) | 295
percentage of participants
  ST Elevation Sensitivity | 100 [100 to 100]
  ST Elevation Specificity | 100 [100 to 100]
  ST Elevation PPV | 100 [100 to 100]
  ST Elevation NPV | 100 [100 to 100]
  ST Depression Sensitivity | 100 [100 to 100]
  ST Depression Specificity | 100 [100 to 100]
  ST Depression PPV | 100 [100 to 100]
  ST Depression NPV | 100 [100 to 100]
  T Wave Inversion Sensitivity | 95 [92 to 97]
  T Wave Inversion Specificity | 80 [68 to 92]
  T Wave Inversion PPV | 97 [95 to 99]
  T Wave Inversion NPV | 70 [56 to 83]

2. Primary Outcome: Kappa Agreement Between Synthesized and Actual 18-lead ECGs in the Identification of ST Elevation, ST Depression, and T Wave Inversion
Description: Kappa value for comparison of actual 18-lead ECG vs synthesized ECG leads. All measures at 95% confidence Index.
Time Frame: 30 minutes
Measure: Number (95% Confidence Interval); unit: Kappa
Arm/Group | All Participants
Number analyzed (Participants) | 295
Kappa
  ST Elevation | 1.00 [1.00 to 1.00]
  ST Depression | 1.00 [1.00 to 1.00]
  T Wave Inversion | 0.70 [0.58 to 0.82]

ADVERSE EVENTS:
Time Frame: 30 minutes
Description: All adverse events (all cause mortality, serious-adverse, other - not serious) reported to P.I. in written form via data collection form.
Arm/Group | Test
All-Cause Mortality (participants affected / at risk) | 0/314
Serious Adverse Events (participants affected / at risk) | 0/314
Other Adverse Events (participants affected / at risk) | 0/314

LIMITATIONS AND CAVEATS:
Original goal of 300 subjects was not reached. However, analysis of 295 subjects still yielded statistical valid results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT03426436/Prot_SAP_000.pdf